CLINICAL TRIAL: NCT01221311
Title: Use of Fully-covered, Self-expandable Metallic Stents for First-line Treatment of Benign Bile Duct Strictures
Brief Title: Covered Metallic Stents for First-Line Treatment of Benign Bile Duct Strictures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Gregory A. Cote, Associate Professor of Medicine, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G100118; R21DK090708 (NIH); NCT01432808 (obsolete NCT alias)
Record Dates: First submitted 2010-10-08; First posted 2010-10-15 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Common Bile Duct Stricture
Keywords: stenosis; bile duct; chronic pancreatitis; postoperative; post-liver transplant
MeSH Terms: conditions — Constriction, Pathologic; Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fully Covered Metallic Stent (Experimental): Among patients randomized to the covered, self-expandable metallic stent (cSEMS) group, the endoscopist will deploy a cSEMS of sufficient length to traverse the papilla. Dilation will not be performed unless the cSEMS deployment catheter cannot be advanced over a guidewire beyond the stricture. A biliary sphincterotomy may be performed at the discretion of the treating endoscopist.
  Interventions: Device: Fully covered Metallic Stent
- Plastic Stent (Active Comparator): Patients randomized to the plastic stent (PS) group will be treated using a standard algorithm. Specifically, the stricture will be dilated using a passage dilator and/or dilation balloon catheter, and multiple (as many as technically feasible) PS will be deployed depending on the baseline characteristics of the stricture as well as the diameter of the proximal and distal bile duct (standard of care). The endoscopist will sequentially dilate and upsize the cumulative stent diameter on ensuing endoscopic retrograde cholangiopancreatography (ERCP), until the stricture has been obliterated using clinical and fluoroscopic criteria (details below).
  Interventions: Device: Plastic Stent

INTERVENTIONS:
Device: Fully covered Metallic Stent — Covered Wallflex Biliary (TM)
  Arms: Fully Covered Metallic Stent
Device: Plastic Stent — Patients randomized to the PS group will be treated using a standard algorithm. Specifically, the stricture will be dilated using a passage dilator and/or dilation balloon catheter, and one or two PS will be deployed depending on the baseline characteristics of the stricture as well as the diameter of the proximal and distal bile duct (standard of care). The endoscopist will sequentially dilate and upsize the cumulative stent diameter on ensuing ERCPs, until the stricture has been obliterated using clinical and fluoroscopic criteria.
  Other Names: Polyethylene Stent
  Arms: Plastic Stent

SUMMARY:
The current standard of care for benign bile duct strictures involves placement of multiple plastic stents under endoscopic and fluoroscopic guidance to progressively dilate or stretch it open. This approach necessitates multiple procedures which may extend over one year before the stricture is adequately dilated. The investigators propose a study comparing the standard approach of plastic stenting with the use of newer, fully coated metallic stents which are self-expandable, thereby permitting successful dilation of benign bile duct strictures with fewer procedures.

DETAILED DESCRIPTION:
Randomization, as detailed below, is stratified by etiology of the stricture: chronic pancreatitis and postoperative (such as post-liver transplant).

ELIGIBILITY:
Inclusion Criteria:

* Bismuth Type I benign bile duct stricture
* Objective signs/symptoms related to the stricture

Exclusion Criteria:

* Suspected malignant etiology for the stricture
* Prior endotherapy within one year of presentation,except in the following two scenarios: 1) Early (< 30 days) stent placement following liver transplant; 2) in patients with chronic pancreatitis, single plastic stent placed during presenting ERCP while evaluating for malignancy
* Bismuth Type II-IV stricture
* Proximal common hepatic duct diameter < 6 mm
* Intact gallbladder, except in cases where a stent can be deployed > 1cm below the cystic duct insertion
* Age < 18 years, pregnancy, incarceration, inability to provide informed consent
* Karnofsky score ≤ 40
* Inability to pass a guidewire proximal to the stricture
* Stricture > 8cm in length
* Life expectancy < 1 year
* Concomitant nonanastomotic biliary strictures or biliary casts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-01; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Cote, MD, MS, Principal Investigator — Medical University of South Carolina
Locations (8):
- United States (7):
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Digestive Health Associates of Texas, Dallas, Texas
- Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cote GA, Slivka A, Tarnasky P, Mullady DK, Elmunzer BJ, Elta G, Fogel E, Lehman G, McHenry L, Romagnuolo J, Menon S, Siddiqui UD, Watkins J, Lynch S, Denski C, Xu H, Sherman S. Effect of Covered Metallic Stents Compared With Plastic Stents on Benign Biliary Stricture Resolution: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1250-7. doi: 10.1001/jama.2016.2619. PMID 27002446

RESULTS

PARTICIPANT FLOW:
Groups:
- Plastic Stent: Patients randomized to the plastic stent (PS) group will be treated using a standard algorithm. Specifically, the stricture will be dilated using a passage dilator and/or dilation balloon catheter, and multiple (as many as technically feasible) PS will be deployed depending on the baseline characteristics of the stricture as well as the diameter of the proximal and distal bile duct (standard of care). The endoscopist will sequentially dilate and upsize the cumulative stent diameter on ensuing endoscopic retrograde cholangiopancreatography (ERCP), until the stricture has been obliterated using clinical and fluoroscopic criteria (details below).
  Plastic Stent: Patients randomized to the PS group will be treated using a standard algorithm. Specifically, the stricture will be dilated using a passage dilator and/or dilation balloon catheter, and one or two PS will be deployed depending on the baseline characteristics of the stricture as well as the diameter of the proximal and distal
Period: Overall Study
Arm/Group | Fully Covered Metallic Stent | Plastic Stent
Started | 57 | 55
Completed | 57 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Plastic Stent: Patients randomized to the plastic stent (PS) group will be treated using a standard algorithm. Specifically, the stricture will be dilated using a passage dilator and/or dilation balloon catheter, and multiple (as many as technically feasible) PS will be deployed depending on the baseline characteristics of the stricture as well as the diameter of the proximal and distal bile duct (standard of care). The endoscopist will sequentially dilate and upsize the cumulative stent diameter on ensuing endoscopic retrograde cholangiopancreatography (ERCP), until the stricture has been obliterated using clinical and fluoroscopic criteria.
- Total: Total of all reporting groups
Arm/Group | Fully Covered Metallic Stent | Plastic Stent | Total
Number analyzed (Participants) | 57 | 55 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.4) | 56.7 (11) | 55.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 38 | 38 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Early Clinical Success
Description: Early clinical success will be defined as fluoroscopic resolution at the time all stent(s) are removed. If there is a persistent stricture after 12 months of stent therapy in either group, the patient will be classified as a clinical failure. We will compare early clinical success rates in each group.
Time Frame: Post-stent removal (up to one year after enrollment)
Population: The number of participants analyzed is lower than the number of patients randomized, due to patients who dropped out of the study before all stents were removed.
Measure: Count of Participants; unit: Participants
Arm/Group | Fully Covered Metallic Stent | Plastic Stent
Number analyzed (Participants) | 54 | 48
Participants | 50 | 41

ADVERSE EVENTS:
Arm/Group | Fully Covered Metallic Stent | Plastic Stent
Serious Adverse Events (participants affected / at risk) | 14/57 | 9/55
Other Adverse Events (participants affected / at risk) | 8/57 | 8/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fully Covered Metallic Stent (N=57) | Plastic Stent (N=55)
Stent migration (Gastrointestinal disorders) | 14 (16) | 9 (10)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fully Covered Metallic Stent (N=57) | Plastic Stent (N=55)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No